CLINICAL TRIAL: NCT07285356
Title: GLOX-PEN: Phase II Clinical Trial to Evaluate the Use of Surgical Gloves for the Prevention of Oxaliplatin-Induced Peripheral Neuropathy
Brief Title: Study to Evaluate the Use of Surgical Gloves for the Prevention of Oxaliplatin-Induced Peripheral Neuropathy
Acronym: GLOX-PEN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AC Camargo Cancer Center (Other)
Collaborators: Hospital do Cancer de Londrina (Unknown)
Responsible Party: Principal Investigator, Virgilio Souza e Silva, Doctor and Head Oncologist of the Clinical Oncology Department at AC Camargo Cancer Center, AC Camargo Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 90669425.4.1001.5432
Record Dates: First submitted 2025-11-17; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Colon Cancer; Oxaliplatin-induced Peripheral Neuropathy
Keywords: oxaliplatin-induced peripheral neuropathy; Peripheral Neuropathy; Oxaliplatin; Surgical Gloves; Body Mass Index (BMI); Sarcopenia
MeSH Terms: conditions — Colonic Neoplasms; Peripheral Nervous System Diseases; Sarcopenia | interventions — Gloves, Surgical

STUDY DESIGN:
Intervention Model Description: This study is a prospective, open-label, randomized, controlled, multicenter clinical trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgical Gloves (Experimental): During each chemotherapy cycle, patients in the experimental arm will wear compressive surgical gloves (0.5 size smaller than recommended based on palmar surface measurement) on both hands, which will be put on 30 minutes before the infusion and remain in place until 30 minutes after the end of the chemotherapy infusion.
  Interventions: Device: Surgical Gloves
- No Surgical Gloves (No Intervention): The control arm will receive treatment according to current recommendations without the use of any devices on the hands.

INTERVENTIONS:
Device: Surgical Gloves — During each chemotherapy cycle, patients in the experimental group will wear compressive surgical gloves (one size smaller than recommended based on palmar surface measurement) on both hands, which will be put on 30 minutes before the infusion and remain in place until 30 minutes after the end of the chemotherapy infusion.
  Arms: Surgical Gloves

SUMMARY:
The primary objective of this randomized clinical trial is to assess whether the use of surgical gloves during treatment can prevent the occurrence of oxaliplatin-induced peripheral neuropathy.

DETAILED DESCRIPTION:
Gastrointestinal tumors account for one-quarter of the global cancer incidence and one-third of cancer-related deaths. Chemotherapy-induced peripheral neuropathy (CIPN) is a common adverse effect of oxaliplatin-based treatments. CIPN can lead to an extremely painful and debilitating process, causing significant loss of functional abilities and negatively affecting the quality of life of these patients, as well as activities of daily living (ADLs) such as walking, buttoning clothes, writing, brushing teeth, among others. This condition can even result in a state of vulnerability, with a high risk of falls and other injuries.

Primary Objective and Study Rationale:

Oxaliplatin, widely used to treat patients with colorectal neoplasms, is associated with chemotherapy-induced peripheral neuropathy (CIPN). Given the high prevalence and negative impact of CIPN on quality of life and adherence to cancer treatment, there is a significant gap in identifying effective prevention and management strategies. Although recent evidence suggests that surgical gloves (SG) can mitigate paclitaxel-induced peripheral neuropathy, SGs have not been tested for the prevention of oxaliplatin-induced peripheral neuropathy (OIPN). Therefore, the primary objective of this randomized clinical trial is to evaluate whether the use of SGs during treatment can prevent the occurrence of grade 2 or higher OIPN in the hands, as assessed by CTCAE v5.0 and PRO-CTCAE.

Secondary Objective:

To determine the relationship between Body Mass Index and the presence of sarcopenia, with the occurrence of OIPN; To evaluate the impact of OIPN on patients' health-related quality of life (HRQoL) using the EORTC QLQ-C30 questionnaire; To assess symptoms and functional limitations associated with OIPN using the EORTC QLQ-CIPN20 questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older who have provided written informed consent.
* Colon adenocarcinoma with high-risk stage III (pT4pN2) or stage IV.
* Oxaliplatin-based treatment in the context of localized or metastatic disease.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.

Exclusion Criteria:

* Pre-existing neuropathy.
* Uncontrolled diabetes.
* known glove allergies.
* Prior treatment with paclitaxel, docetaxel or oxaliplatin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-10-06 (Actual); Primary Completion 2026-09-18 (Estimated); Study Completion 2026-09-18 (Estimated)

PRIMARY OUTCOMES:
Oxaliplatin-Induced Peripheral Neuropathy | Baseline, 2 months, 4 months and 6 months
  The primary objective of this randomized clinical trial is to evaluate whether the use of surgical gloves during treatment can prevent the occurrence of grade 2 or higher oxaliplatin-induced peripheral neuropathy in the hands, as assessed by CTCAE v5.0 .

SECONDARY OUTCOMES:
Sarcopenia assessing by muscle strength, muscle quantity/quality, and physical performance, Body Mass Index (BMI) evaluated by a mathematical formula (kg/m2). | Baseline, 2 months, 4 months and 6 months
  To determine the relationship between BMI and the presence of sarcopenia, with the occurrence of oxaliplatin-induced peripheral neuropathy (OIPN);
Health-related Quality of life questionaries | Baseline, 2 months, 4 months and 6 months
  To evaluate the impact of OIPN on patients' health-related quality of life (HRQoL) using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire - Core 30 (EORTC QLQ-C30). For the Functional Scales, higher scores indicate better functioning (0=poorest ; 100=best). For the Symptom Scales, higher scores indicate greater symptom severity (0=no symptoms; 100=severe). For the Global Health Status/Quality of Life Scale, higher scores reflect a better overall perception of health and quality of life (0=poorest; 100=best).
Functional limitations associated with OIPN | Baseline, 2 months, 4 months and 6 months
  To assess symptoms and functional limitations associated with OIPN using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-CIPN20). All scores are transformed into a standardized 0-100 scale, with higher scores indicating severe symptoms.
Patient reported Peripheral Neuropathy | Baseline, 2 months, 4 months and 6 months
  Patient reported Oxaliplatin-Induced Peripheral Neuropathy assessed by PRO- CTCAE.

CONTACTS AND LOCATIONS:
Overall Officials: Bruna Catin Kupper, Nurse, PhD, Study Chair — AC Camarco Cancer Center; Éverton Germano Melo, Medical Doctor, Principal Investigator — Londrina Cancer Hospital; Virgilio Souza Silva, Medical Doctor, PhD, Principal Investigator — AC Camargo Cancer Center; Karina Oliveira Ribeiro, Nurse, Study Chair — AC Camargo Cancer Center
Locations (1):
- A.C. Camargo Cancer Center, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Incidence of grade 2 or higher oxaliplatin-induced peripheral neuropathy (OIPN) in the hands, as assessed by CTCAE v5.0.; Proportion of patients requiring dose adjustments and/or treatment interruptions; Grade 2 or higher OIPN in the patients' feet; Health-related quality of life (HRQoL) using the EORTC QLQ-C30 questionnaire; Assessment of symptoms and associated functional limitations due to OIPN using the EORTC QLQ-CIPN20 questionnaire; Evaluation of the correlation between body mass index (BMI) and the presence of sarcopenia, with the occurrence of OIPN.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Start date: October 2025 End date: September 2026
Access Criteria: All Principal Investigators and Chairs of this trial
URL: https://accamargo.org.br/pacientes/estudos-clinicos/lista-de-estudos-clinicos

REFERENCES:
- [Background] Smith EM. Current methods for the assessment and management of taxane-related neuropathy. Clin J Oncol Nurs. 2013 Feb;17 Suppl:22-34. doi: 10.1188/13.CJON.S1.22-34. PMID 23360700
- [Background] Soveri LM, Lamminmaki A, Hanninen UA, Karhunen M, Bono P, Osterlund P. Long-term neuropathy and quality of life in colorectal cancer patients treated with oxaliplatin containing adjuvant chemotherapy. Acta Oncol. 2019 Apr;58(4):398-406. doi: 10.1080/0284186X.2018.1556804. Epub 2019 Jan 14. PMID 30638100
- [Background] Tofthagen C. Patient perceptions associated with chemotherapy-induced peripheral neuropathy. Clin J Oncol Nurs. 2010 Jun;14(3):E22-8. doi: 10.1188/10.CJON.E22-E28. PMID 20529785
- [Background] Wang S, Zheng R, Li J, Zeng H, Li L, Chen R, Sun K, Han B, Bray F, Wei W, He J. Global, regional, and national lifetime risks of developing and dying from gastrointestinal cancers in 185 countries: a population-based systematic analysis of GLOBOCAN. Lancet Gastroenterol Hepatol. 2024 Mar;9(3):229-237. doi: 10.1016/S2468-1253(23)00366-7. Epub 2024 Jan 4. PMID 38185129